CLINICAL TRIAL: NCT06529705
Title: Performance and Safety Evaluation of the EkiYou V2 Application in Patients With Diabetes Using Multiple Daily Insulin Injections (EkiYou-Study1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: DiappyMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0453; 2024-A00433-44 (Other: ANSM)
Record Dates: First submitted 2024-07-15; First posted 2024-07-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Type 1; Diabetes Type 2 on Insulin; Pancreatogenous Diabetes
Keywords: Decision support system; Digital health; Continuous glucose monitoring; Precision insulin management; Insulin titration
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Adults with type 1, type 2 diabetes or pancreatogenic diabetes treated by multiple daily insulin injections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with diabetes treated by MDI (Experimental)
  Interventions: Device: EkiYou V2

INTERVENTIONS:
Device: EkiYou V2 — Use of a mobile application that help users to evaluate their daily bolus and basal insulin needs, and that adjusts at weekly basis their insulin to carb ratios, correction factor and basal dose.

SUMMARY:
EkiYou-Study-1 is an interventional before/after clinical investigation according to EU 2017/745. It is conducted in 21 adults with diabetes and treated by multiple daily insulin injections.

After a run-in period of 2 weeks, participants will receive for 6 weeks EkiYou V2 application that will help them to estimate their daily bolus and basal insulin doses. This device weekly adjusts insulin parameters including : basal insulin dose, insulin to carb ratios and correction factor.

The aim of the study is to assess the safety and performance of EkiYou V2 device. Data on glycemic control, safety, quality of life and satisfaction of participants will be collected.

DETAILED DESCRIPTION:
Participants of the study must be adults treated by multiple daily insulin injection in a basal/bolus insulin schema and users of a continuous glucose monitor (CGM). The study involves 5 visits, each two weeks. Participants will be included for 8 weeks divided in two distinct periods :

* Run-in period for two weeks to collect glycemic control at baseline with their standard insulin management
* Intervention period for 6 weeks where participant will receive the investigational device EkiYou V2 to manage their insulin injection.

EkiYou V2 device is a new version of the previously CE-Marked device EkiYou V1. It is a decision support that include the following features to participants:

* Carbohydrate counting through an extensive food database with more than 200k items.
* Bolus calculation based on their meal, physical activity and blood glucose.
* Bolus correction advice.
* Long-acting insulin reminders and automatic periodic titration.
* Insulin-to-carb ratios and correction factor automatic adjustment.

ELIGIBILITY:
Inclusion Criteria :

* Be over 18 years old;
* Have type 1, type 2, or pancreatogenic diabetes;
* Have been treated with multiple daily injections of insulin in a basal/bolus regimen for at least 6 months;
* Be using a continuous glucose monitoring device such as Dexcom G6, Dexcom One or Freestyle Libre for at least 2 weeks;
* Have a time in the glycemic target range (70-180 mg/dl) of less than 70%;
* Require at least 15 units of insulin therapy per day;
* Use a rapid-acting insulin compatible with the device, such as Novorapid, Humalog, Apidra, Asparte, Sanofi, Fiasp, or Lyumjev;
* Use a long-acting insulin compatible with the device, such as Lantus, Abasaglar, Toujeo, Levemir, or Tresiba;
* Be able to read and use a smartphone;
* Have no visual impairment requiring a specific font for smartphones;
* Have basic knowledge of smartphone use;
* Indicate their willingness to follow the protocol and sign a written informed consent

Exclusion Criteria:

* Ketoacidosis or severe level 3 hypoglycemia requiring third-party intervention within 6 months prior to inclusion;
* Treatment with any hypoglycemia-inducing agent other than insulin (including sulfonylureas and SGLT-2 inhibitors);
* Daily insulin requirement exceeding 200 U/day;
* Suffering from gastroparesis;
* Pancreatopathy secondary to chronic alcoholism;
* Known medical condition that, in the investigator's opinion, may interfere with the protocol;
* Participation in another clinical trial or administration of an unapproved medication within 4 weeks prior to screening;
* Not affiliated with a social security system;
* Vulnerable subject: minors, or adults under protection as defined by the Public Health Code, pregnant or breastfeeding women, subjects under guardianship or deprived of liberty;
* Person under legal protection;
* Person participating in another study with an ongoing exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of time in range 70-180 mg/dL | Through study completion, an average of 8 weeks
  Time in range is the amount of time spent in the target glucose range-between 70 and 180 mg/dL-as measured by CGM

SECONDARY OUTCOMES:
Number of non-serious adverse events related or unrelated to the device | Through study completion, an average of 8 weeks
  Severe hypoglycemia (Level 3) with blood glucose below 54 mg/dL and requiring assistance from an external person for carbohydrates intake or glucagon use.
Number of non-serious adverse events related or unrelated to the device | Through study completion, an average of 8 weeks
  Severe hyperglycemia (Level 3) defined by the presence of ketonemia > 3 mmol/L or ketonemia > 1 mmol/L and requiring consultation with a healthcare professional.
Number of serious clinical adverse events (SAEs) | Through study completion, an average of 8 weeks
  Number of severe level 3 hypoglycemic events requiring hospitalization
Number of serious clinical adverse events (SAEs) | Through study completion, an average of 8 weeks
  Number of episodes of diabetic ketoacidosis requiring hospitalization
Number of other serious adverse events related or unrelated to the device | Through study completion, an average of 8 weeks
Number of non-serious and unexpected adverse events related to the device | Through study completion, an average of 8 weeks
Change in the percentage of time below 54 mg/dL | 2 weeks follow-up
  Percentage of time with glucose below 54 mg/dL as measured by CGM
Change in the percentage of time below 54 mg/dL | 8 weeks follow-up
  Percentage of time with glucose below 54 mg/dL as measured by CGM
Change in the percentage of time below 70 mg/dL | 2 weeks follow-up
  Percentage of time with glucose below 70 mg/dL as measured by CGM
Change in the percentage of time below 70 mg/dL | 8 weeks follow-up
  Percentage of time with glucose below 70 mg/dL as measured by CGM
Change in the percentage of time above 180 mg/dL | 2 weeks follow-up
  Percentage of time with glucose above 180 mg/dL as measured by CGM
Change in the percentage of time above 180 mg/dL | 8 weeks follow-up
  Percentage of time with glucose above 180 mg/dL as measured by CGM
Change in the percentage of time above 250 mg/dL | 2 weeks follow-up
  Percentage of time with glucose above 250 mg/dL as measured by CGM
Change in the percentage of time above 250 mg/dL | 8 weeks follow-up
  Percentage of time with glucose above 250 mg/dL as measured by CGM
Change in the Glucose Management Indicator (GMI) | 2 weeks follow-up
  GMI as measured by CGM
Change in the Glucose Management Indicator (GMI) | 8 weeks follow-up
  GMI as measured by CGM
Percentage of patients with time in range 70-180 mg/dL above or equal to 70% | 2 weeks follow-up
  Time in range 70-180 mg/dL as measured by CGM
Percentage of patients with time in range 70-180 mg/dL above or equal to 70% | 8 weeks follow-up
  Time in range 70-180 mg/dL as measured by CGM
Change in Mean blood glucose level | 2 weeks follow-up
  Mean sensor glucose as measured by CGM
Change in Mean blood glucose level | 8 weeks follow-up
  Mean sensor glucose as measured by CGM
Change in Coefficient of variation of blood glucose | 2 weeks follow-up
  Coefficient of variation of blood glucose as measured by CGM
Change in Coefficient of variation of blood glucose | 8 weeks follow-up
  Coefficient of variation of blood glucose as measured by CGM
Number of level 2 hypoglycemic episodes | 2 weeks follow-up
  Defined as blood glucose below 54 mg/dL for more than 15 minutes
Number of level 2 hypoglycemic episodes | 8 weeks follow-up
  Defined as blood glucose below 54 mg/dL for more than 15 minutes
Total Daily Insulin (Units/kg) | 2 weeks follow-up
Change in Total Daily Insulin (Units/kg) | 8 weeks follow-up
Total Insulin Delivered Via Basal (Units/kg) | 2 weeks follow-up
Change in total Insulin Delivered Via Basal (Units/kg) | 8 weeks follow-up
Number per day and total Insulin Delivered Via Bolus (Units/kg) | 2 weeks follow-up
Change in number per day and total Insulin Delivered Via Bolus (Units/kg) | 8 weeks follow-up
Number of connectivity issues with the application reported by the user | 8 weeks follow-up
Questionnaire System Usability scale | 8 weeks follow-up
  Device usability questionnaire. The lower the score, more the participant agrees with the item; a higher score indicates disagreement with the item.
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | At inclusion visit
  Quality of life associated with diabetes questionnaire. Treatment Satisfaction: Items 1, 4, 5, 6, 7 & 8 are summed to produce a Treatment Satisfaction score (range: 0 to 36). The higher the score, the greater the satisfaction with treatment.
  Individual satisfaction with treatment items (items 1, 4, 5, 6, 7 & 8) can be considered separately: All rated: 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied, inconvenient, inflexible, etc.). The higher the score, the greater the satisfaction with each aspect of treatment.
  'Perceived frequency of hyperglycaemia' (item 2) & 'Perceived frequency of hypoglycaemia' (item 3): Both rated: 6 ('most of the time') to 0 ('none of the time'). Here, lower scores indicate blood glucose levels closer to the ideal. Higher scores indicate problems
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 8 weeks follow-up
  Quality of life associated with diabetes questionnaire Treatment Satisfaction: Items 1, 4, 5, 6, 7 & 8 are summed to produce a Treatment Satisfaction score (range: 0 to 36). The higher the score, the greater the satisfaction with treatment.
  Individual satisfaction with treatment items (items 1, 4, 5, 6, 7 & 8) can be considered separately: All rated: 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied, inconvenient, inflexible, etc.). The higher the score, the greater the satisfaction with each aspect of treatment.
  'Perceived frequency of hyperglycaemia' (item 2) & 'Perceived frequency of hypoglycaemia' (item 3): Both rated: 6 ('most of the time') to 0 ('none of the time'). Here, lower scores indicate blood glucose levels closer to the ideal. Higher scores indicate problems
Hypoglycemia Fear Survey 2 (HFS II) | At inclusion visit
  Fear of hypoglycemia questionnaire. Behavioral Subscale, Items: 1-15 Score Range: 0 to 75. Higher scores indicate more frequent behaviors aimed at avoiding hypoglycemia, reflecting a greater fear of low blood sugar episodes.
  Worry Subscale, Items: 16-33 Score Range: 0 to 90. Higher scores suggest greater concern or anxiety about the consequences of hypoglycemia, including physical symptoms and impact on daily activities.
  Total Score Range: 0 to 165 (sum of both subscales). A higher total score indicates a more intense overall fear of hypoglycemia, affecting both behavior and emotional well-being.
Hypoglycemia Fear Survey 2 (HFS II) | 8 weeks follow-up
  Fear of hypoglycemia questionnaire. Behavioral Subscale, Items: 1-15 Score Range: 0 to 75. Higher scores indicate more frequent behaviors aimed at avoiding hypoglycemia, reflecting a greater fear of low blood sugar episodes.
  Worry Subscale, Items: 16-33 Score Range: 0 to 90. Higher scores suggest greater concern or anxiety about the consequences of hypoglycemia, including physical symptoms and impact on daily activities.
  Total Score Range: 0 to 165 (sum of both subscales). A higher total score indicates a more intense overall fear of hypoglycemia, affecting both behavior and emotional well-being.
Number of daily insulin injections calculated from application data | 8 weeks follow-up
Average number of daily interactions calculated from application data | 8 weeks follow-up
Number of active application users | 8 weeks follow-up
  Defined as at least 14 recorded injections in the application over a 2-week period

CONTACTS AND LOCATIONS:
Overall Officials: Orianne VILLARD, MD, Principal Investigator — CHU de Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France, France